CLINICAL TRIAL: NCT03899636
Title: A Randomized, Multicenter, Controlled, Unblinded Study to Assess the Safety and Efficacy of the NanoKnife® System for the Ablation of Unresectable Stage 3 Pancreatic Adenocarcinoma
Brief Title: A Pivotal Study of Safety and Effectiveness of NanoKnife IRE for Stage 3 Pancreatic Cancer
Acronym: DIRECT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28-001-ONC
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Stage III Pancreatic Cancer
Keywords: Pancreas Cancer; Pancreatic Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Advanced Pancreatic Cancer; Carcinoma, Pancreatic Ductal; Locally Advanced Pancreatic Cancer; Cancer of Pancreas; Pancreatic Tumor; Pancreatic Carcinoma; Unresectable Pancreatic Cancer; LAPC
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- IRE (Experimental)
  Interventions: Drug: Modified FOLFIRINOX Regimen; Device: NanoKnife System
- Control (Active Comparator)
  Interventions: Drug: Modified FOLFIRINOX Regimen

INTERVENTIONS:
Drug: Modified FOLFIRINOX Regimen — Chemotherapy regimen of leucovorin, fluorouracil, irinotecan, and oxaliplatin
Device: NanoKnife System — IRE using NanoKnife System
  Arms: IRE

SUMMARY:
Subjects will be offered the opportunity to participate in a randomized, controlled, 2-arm, unblinded multicenter trial (RCT). There will be 2 study arms: the control arm receiving chemotherapy with the modified FOLFIRINOX regimen alone; and the irreversible electroporation (IRE) arm, receiving chemotherapy with the modified FOLFIRINOX regimen followed by IRE with the NanoKnife System using either an open or a percutaneous approach. All subjects will be treated with the modified FOLFIRINOX regimen for at least 3 months; randomization to either control or IRE arm will take place at the time of completion of the 3 month modified FOLFIRINOX chemotherapy regimen. Randomization will be conducted centrally. Subjects will be randomized in a 1:1 ratio and must be found to have no evidence of disease progression after completion of the 3 month modified FOLFIRINOX chemotherapy regimen in order to participate in the RCT. All radiologic assessments will be performed as consistent with the imaging protocol. All post induction and post IRE treatments are left to the discretion of the treating physician. The minimum period of follow-up will be for 24 months or until death.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Subject is 18 years of age and older.
3. Subject has a diagnosis of unresectable Stage 3 pancreatic adenocarcinoma cancer cytologically or pathologically confirmed per American Joint Committee on Cancer (AJCC) staging criteria.
4. Subject has a tumor evaluated as Stage 3 according to National Comprehensive Cancer Network (NCCN) guidelines, based on radiographic imaging or exploratory surgery.
5. Maximum axial and anterior to posterior tumor dimension of ≤3.5cm, after receiving three months of treatment with the modified FOLFIRINOX regimen.
6. Subject has received 3 months of treatment with the modified FOLFIRINOX regimen.
7. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Subject has an American Society of Anesthesiologists (ASA) classification of physical health status of 1 or 2.

Exclusion Criteria:

1. Subjects who are or may be pregnant as determined by a positive pregnancy test or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 6 months after the last dose of chemotherapy.
2. Subjects who are unable to tolerate general anesthetic with full skeletal muscle blockade.
3. Subjects who are actively bleeding, anticoagulated, coagulopathy, or have any of the following hematology results: hemoglobin less than 10 g/dL without the support of growth factors or transfusions absolute neutrophil count less than 1500 cells/mL; or platelet count less than 100,000.
4. Subjects with the presence of implanted cardiac pacemakers, defibrillators, electronic devices or implanted devices with metal parts in the thoracic cavity at the time of IRE.
5. Subjects with history of epilepsy or other neurological disease.
6. Subjects with renal, cardiac, liver, or hematological abnormalities of concern to the investigator.
7. Subjects with Stage 3, 4, or 5 chronic kidney disease.
8. Subjects receiving IRE for margin accentuation.
9. Subjects who at 3 months after FOLFIRINOX treatment have evidence of disease progression.
10. Participation in another interventional trial for pancreatic cancer.
11. Subjects who did not meet study defined criteria for adequacy of induction treatment at the end of the 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Time (in months) from randomization to the date of death for any reason, assessed through at least 24 months.
  Time (in months) from randomization to the date of death for any reason

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Miami Cancer Institute, Miami, Florida
  - University of South Florida/Tampa, Tampa, Florida
  - Northwest Community Healthcare, Arlington Heights, Illinois
  - Norton Healthcare, Louisville, Kentucky
  - St. Luke's Cancer Center, Easton, Pennsylvania
  - University of Texas-Southwestern, Dallas, Texas

REFERENCES:
- [Derived] Narayanan G, Bilimoria MM, Hosein PJ, Su Z, Mortimer KM, Martin RCG 2nd. Multicenter randomized controlled trial and registry study to assess the safety and efficacy of the NanoKnife(R) system for the ablation of stage 3 pancreatic adenocarcinoma: overview of study protocols. BMC Cancer. 2021 Jul 7;21(1):785. doi: 10.1186/s12885-021-08474-4. PMID 34233640